CLINICAL TRIAL: NCT01459627
Title: Prospective, Randomized, Open Label Trial of 6 Months vs. 12 Months Dual Antiplatelet Therapy After Drug-Eluting Stent Implantation In ST-elevation Myocardial Infarction
Brief Title: Randomized, Open Label Trial of 6 Months Versus 12 Months DAPT After Drug-Eluting Stent in STEMI
Acronym: DAPT-STEMI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maasstad Hospital (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAPT-STEMI
Record Dates: First submitted 2011-10-18; First posted 2011-10-25 (Estimated); Last update posted 2017-09-07 (Actual); Status verified 2017-09

CONDITIONS: Myocardial Infarction; Cardiovascular Disease
Keywords: DAPT- Dual Antiplatelet Therapy; STEMI
MeSH Terms: conditions — Myocardial Infarction; Cardiovascular Diseases; ST Elevation Myocardial Infarction | interventions — 2'-deoxythymidylyl-(3'-5')-2'-deoxyadenosine; Ticagrelor; Prasugrel Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 6 months DAPT (Active Comparator): Dual antiplatelet therapy consisting of aspirin (ASA) and prasugrel or ticagrelor will be discontinued after randomisation.
  Interventions: Other: 6 months DAPT
- 12 months DAPT (Active Comparator): Dual antiplatelet therapy consisting of aspirin (ASA) and prasugrel or ticagrelor will be continued till 12 months after enrollment in the study
  Interventions: Other: 12 months DAPT

INTERVENTIONS:
Other: 6 months DAPT — Dual antiplatelet therapy will be stopped at randomisation to the 6 months DAPT group. Patients will be treated from 6 months onwards only with ASA.
  Other Names: ticagrelor, prasugrel, ASA
  Arms: 6 months DAPT
Other: 12 months DAPT — Dual antiplatelet therapy will be continued till 12 months after enrollment in the study
  Other Names: ticagrelor, prasugrel, ASA
  Arms: 12 months DAPT

SUMMARY:
OBJECTIVE OF THE STUDY: To test the hypothesis that 6 months DAPT (Dual anti-platelet therapy) after second generation DES (Drug Eluting Stent) implantation in STEMI (ST elevation Myocardial Infarction) is not inferior to 12 months DAPT in terms of clinical outcomes (composite endpoint of all-cause mortality, any MI, any revascularization, stroke and major bleeding at 18 months after randomization).

The trial will incorporate two registers studying respectively the safety outcomes of Bivalirudin and Prasugrel combination and Bivalirudin and Ticagrelor combination at 2 and 30 days. Finally the trial design permits assessment of the clinical outcomes after primary PCI for treatment of STEMI with the new Resolute Integrity (Medtronic Santa Rosa Ca, USA) stent at 30 days and 6 months.

DETAILED DESCRIPTION:
BACKGROUND OF THE STUDY: First generation DES (Drug Eluting Stents) have significantly reduced the restenosis rates compared to the BMS (Bare Metal Stents) but have raised concerns regarding higher rates and ongoing propensity for stent thrombosis. Based on these concerns current guidelines advocate dual antiplatelet therapy (DAPT, aspirin plus P2Y12 inhibitor) to be continued for up to 1 year after DES implantation. Large registries analyzing recent data now challenge these recommendations and suggest no increase in mortality or (late) stent thrombosis when DAPT is discontinued after 6 months.

STUDY DESIGN: This is a prospective, randomized, open-label trial testing the hypothesis that 6 months DAPT after second generation drug eluting stent (DES) implantation in STEMI is not inferior to 12 months DAPT in terms of clinical outcomes. Patients with STEMI undergoing primary PCI will be enrolled at presentation. Only those patients who are event-free (death, MI, ST, TVR/TLR or unscheduled revascularization with DES in the first 6 months and stroke or bleeding requiring discontinuation of DAPT) and on DAPT at 6 months after primary PCI will be randomized (1:1 fashion) between single (aspirin) versus dual antiplatelet therapy (aspirin plus P2Y12) for an additional 6 months (up to 12 months after primary PCI) and assessed at 18 months post randomization.

STUDY POPULATION: Patients between 18 and 85 years, presenting with STEMI undergoing PCI with DES implantation.

INTERVENTION: Patients, who are event-free and stil on DAPT at 6 months after primary PCI will be randomized (1:1 fashion) between single (aspirin) versus dual antiplatelet therapy (aspirin plus P2Y12) for an additional 6 months (up to 12 months after primary PCI).

PRIMARY STUDY PARAMETERS/OUTCOME OF THE STUDY:

DAPT STEMI trial Composite endpoint of all cause mortality, any MI, any revascularization, stroke, ST and Bleeding (TIMI) (net MACCE) at 18 months after randomization.

Registry Bivalirudin/Prasugrel and Bivalirudin/Ticagrelor All cause mortality, MI, Stroke, ST and bleeding (following BARC) at 2 and 30 days.

Report Resolute Integrity Primary endpoint of DAPT-STEMI, at 30 days and 6 months.

ELIGIBILITY:
Inclusion Criteria:

STEMI patients between 18-85 years who underwent primary PCI with DES implantation.

Exclusion criteria enrolment:

* Intolerance to Aspirin, Prasugrel, Ticagrelor, Heparin, Bivalirudin, Zotarolimus or Everolimus.
* Known bleeding diathesis or known coagulopathy.
* Planned elective surgical procedure necessitating interruption of dual antiplatelet therapy during the first 6 months after randomization.
* History of stent thrombosis
* DES in main left coronary artery
* Active bleeding, known bleeding diathesis or known coagulopathy.
* Planned elective surgical procedure necessitating interruption of dual antiplatelet therapy during the first 6 months after randomization.
* Oral anticoagulant therapy with Coumadin derivates
* Malignancies or other comorbidity with a life expectancy of less than one year or that may result in protocol noncompliance
* Pregnancy (present, suspected or planned) or positive pregnancy test (in women with childbearing potential a negative pregnancy test is mandatory)

Exclusion criteria randomization:

* Occurrence of death, myocardial infarction, stent thrombosis and target vessel or lesion revascularization during the first 6 months after inclusion.
* Stroke or bleeding requiring discontinuation of DAPT during the first 6 months after inclusion.
* Oral anticoagulant therapy

Registry

Exclusion criteria

* Intolerance to Prasugrel, Ticagrelor, Bivalirudin.
* Known bleeding diathesis or known coagulopathy

Report Resolute Integrity Exclusion criteria

• See exclusion criteria enrollment DAPT-STEMI protocol

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2011-12; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Net MACCE | 18 months
  DAPT-STEMI trial: Composite endpoint of all cause mortality, any myocardial infarction (MI) , any revascularization, stroke and major bleeding (TIMI) (net MACCE) at 18 months after randomization

SECONDARY OUTCOMES:
All cause mortality, MI, Stroke, ST and bleeding | 2 days
  Primary outcome of Registry: All cause mortality, MI, Stroke, ST and Bleeding(following BARC)at 2 days.
All cause mortality, MACCE, TIMI | 9 months
  DAPT-STEMI: All cause mortality, any MI, stroke, stent thrombosis (ST) and major bleeding (TIMI) at 9 months after randomization
ST definite/probable | 9 months
  DAPT-STEMI: ST definite/probable academic research consortium (ARC) definition at 9 months post randomization.
all cause mortality | 9 months
  DAPT-STEMI: All cause mortality at 9 months after randomization.
Cardiac mortality | 9 months
  DAPT-STEMI: Cardiac mortality at 9 months after randomization.
MI | 9 months
  DAPT-STEMI: Any MI at 9 months after randomization.
Target vessel MI | 9 months
  DAPT-STEMI: Target vessel MI at 9 months after randomization.
Bleeding | 9 months
  DAPT-STEMI: Bleeding at 9 months after randomization.
stroke | 9 months
  DAPT-STEMI: Stroke at 9 months after randomization.
Target vessel revascularization | 9 months
  DAPT-STEMI: Target vessel revascularization (TVR) at 9 months after randomization.
Target lesion revascularization | 9 months
  DAPT-STEMI: Target lesion revascularization (TLR) at 9 months after randomization.
Target vessel failure | 9 months
  DAPT STEMI: Target vessel failure (TVF) at 9 months after randomization.
Target lesion failure | 9 months
  DAPT-STEMI: Target lesion failure (TLF), at 9 months after randomization.
net MACCE | 30days
  Primary endpoint of Report Resolute Integrity: Composite endpoint of all cause mortality, any myocardial infarction (MI) , any revascularization, stroke and major bleeding (TIMI) (net MACCE) at 30 days after randomization.
  Secondary endpoints of Report Resolute Integrity: Secondary endpoints of DAPT-STEMI at 30 days.
All cause mortality, MI, Stroke, ST and bleeding | 30 days
  Primary outcome of registry: All cause mortality, MI,Stroke, ST and Bleeding (following BARC) at 30 days.
net MACCE | 6 months
  Primary endpoint of Report Resolute Integrity: Composite endpoint of all cause mortality, any myocardial infarction (MI) , any revascularization, stroke and major bleeding (TIMI) (net MACCE) at 6 months after randomization.
  Secondary endpoints of Report Resolute Integrity: Secondary endpoints of DAPT-STEMI at 6 monthss.
All cause mortality, MACCE, TIMI | 18 months
  DAPT-STEMI: All cause mortality, any MI, stroke, stent thrombosis (ST) and major bleeding (TIMI) at 18 months after randomization
ST definite/probable | 18 months
  DAPT-STEMI: ST definite/probable academic research consortium (ARC) definition at 18 months post randomization.
All cause mortality | 18 months
  DAPT-STEMI: All cause mortality at 18 months after randomization.
Cardiac mortality | 18 months
  DAPT-STEMI: Cardiac mortality at 18 months after randomization.
MI | 18 months
  DAPT-STEMI: Any MI at 18 months after randomization.
Target vessel MI | 18 months
  DAPT-STEMI: Target vessel MI at 18 months after randomization.
Bleeding | 18 months
  DAPT-STEMI: Bleeding at 18 months after randomization.
Stroke | 18 months
  DAPT-STEMI: Stroke at 18 months after randomization.
Target vessel revascularization | 18 months
  DAPT-STEMI: Target vessel revascularization (TVR) at 18 months after randomization.
Target lesion revascularization | 18 months
  DAPT-STEMI: Target lesion revascularization (TLR) at 18 months after randomization.
Target vessel failure | 18 months
  DAPT STEMI: Target vessel failure (TVF) at 18 months after randomization.
Target lesion failure | 18 months
  DAPT-STEMI: Target lesion failure (TLF), at 18 months after randomization.
ST following ARC | 2 days
  Registry: ST following ARC definition at 2 days
ST following ARC | 30 days
  Registry: ST following ARC definition at 30 days
All cause mortality | 2 days
  Registry: All cause mortality at 2 days
All cause mortality | 30 days
  Registry: All cause mortality at 30 days
Cardiac mortality | 2 days
  Registry: Cardiac Mortality at 2 days
Cardiac Mortality | 30 days
  Registry: Cardiac Mortality at 30 days
All MI | 2 days
  Registry: All MI at 2 days.
All MI | 30 days
  Registry: All MI at 30 days.
Target vessel MI | 2 days
  Registry: Target vessel MI at 2 days.
Target vessel MI | 30 days
  Registry: Target vessel MI at 30 days.
Bleeding BARC | 2 days
  Registry: Bleeding (BARC) at 2 days
Bleeding (BARC) | 30 days
  Registry: Bleeding (BARC) at 30 days
Stroke | 2 days
  Registry: Stroke at 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Elvin Kedhi, MD PHD, Principal Investigator — Isala; Martin van der Ent, MD PhD, Principal Investigator — Maasstadhospital / MCR B.V.; Clemens von Birgelen, MD PhD, Study Chair — Medisch Spectrum Twente; Felix Zijlstra, MD PhD, Study Chair — Erasmus Medisch Centrum
Locations (16):
- Netherlands (8):
  - VU medisch Centrum, Amsterdam
  - Amphia ziekenhuis, Breda
  - Medisch Spectrum Twente, Enschede
  - Atrium MC Parkstad, Heerlen
  - Maasstadhospital, Rotterdam
  - Erasmus MC, Rotterdam
  - Haga Hospital, The Hague
  - Isala Clinics, Zwolle
- Oslo University Hospital, Oslo, Norway
- Poland (6):
  - Amerykańskie Kliniki Serca, Bielsko-Biala
  - Małopolskie Centrum Sercowo-Naczyniowe PAKS, Chrzanów
  - Polsko-Amerykańskie Kliniki Serca, Dąbrowa Górnicza
  - Polsko_Amerykanskei Kliniki Serca, Kędzierzyn-Koźle
  - University Hospital in Krakow, Krakow
  - Polsko_Amerykanskei Kliniki Serca, Nysa
- Hôpital Cantonal Fribourg, Fribourg, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kedhi E, Delewi R, Fabris E, De Luca G, Hermanides RS, van den Ent M, Buszman P, Zijlstra F, Song YB, Gwon HC, Hahn JY. Duration of dual antiplatelet therapy after myocardial infarction: Insights from a pooled database of the SMART-DATE and DAPT-STEMI trials. Atherosclerosis. 2020 Dec;315:55-61. doi: 10.1016/j.atherosclerosis.2020.11.003. Epub 2020 Nov 9. PMID 33227548
- [Derived] Postma W, Fabris E, Van der Ent M, Hermanides R, Buszman P, Von Birgelen C C, Cook S, Wedel H, De Luca G, Delewi R, Zijlstra F, Kedhi E. Resolute zotarolimus-eluting stent in ST-elevation myocardial infarction (resolute-STEMI): A prespecified prospective register from the DAPT-STEMI trial. Catheter Cardiovasc Interv. 2020 Mar 1;95(4):706-710. doi: 10.1002/ccd.28376. Epub 2019 Jul 3. PMID 31268629
- [Derived] Kedhi E, Fabris E, van der Ent M, Buszman P, von Birgelen C, Roolvink V, Zurakowski A, Schotborgh CE, Hoorntje JCA, Eek CH, Cook S, Togni M, Meuwissen M, van Royen N, van Vliet R, Wedel H, Delewi R, Zijlstra F. Six months versus 12 months dual antiplatelet therapy after drug-eluting stent implantation in ST-elevation myocardial infarction (DAPT-STEMI): randomised, multicentre, non-inferiority trial. BMJ. 2018 Oct 2;363:k3793. doi: 10.1136/bmj.k3793. PMID 30279197